CLINICAL TRIAL: NCT05247268
Title: Gonadotropin-releasing Hormone Agonist Combined With Letrozole Compared With Megestrol Acetate or Medroxyprogesterone Acetate Alone as Fertility-sparing Treatment in Early Endometrial Cancer
Brief Title: Gonadotropin-releasing Hormone Agonist (GnRHa) Plus Letrozole In Young Women With Early Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Prof.Dr., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211032
Record Dates: First submitted 2022-01-16; First posted 2022-02-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Neoplasm Malignant Stage I
Keywords: early endometrial carcinoma; fertility-preserving treatment; gonadotropin-releasing hormone analogue; aromatase inhibitors
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Megestrol Acetate; Tablets; Medroxyprogesterone Acetate; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRHa+letrozole (Experimental): Patients will be stratified into BMI≥28kg/m2 group and BMI<28kg/m2 group. Patients in BMI≥28kg/m2 or BMI<28kg/m2 group will be randomly assigned (1:1) to GnRHa+letrozole group or MA/MPA group. Patients who will be assigned to GnRHa+letrozole group will receive triprorelin acetate (intramuscular injection of 3.75mg was given 4 weeks apart and the maximum use are 6 courses) plus letrozole (2.5mg oral daily and no more than 24 weeks). Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Triprorelin Acetate; Drug: Letrozole 2.5mg
- MA/MPA (Active Comparator): Patients will be stratified into BMI≥28kg/m2 group and BMI<28kg/m2 group. Patients in BMI≥28kg/m2 or BMI<28kg/m2 group were randomly assigned (1:1) to GnRHa+letrozole group or MA/MPA group.Patients assigned to MA/MPA group will receive MA/MPA (160 mg oral MA daily or 500 mg oral MPA daily).Then every 3 months, an hysteroscopy will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol Acetate 160 MG Oral Tablet; Drug: Medroxyprogesterone Acetate 500 MG

INTERVENTIONS:
Drug: Megestrol Acetate 160 MG Oral Tablet — At a dosage of 160 mg/day
  Other Names: Megestrol Acetate
  Arms: MA/MPA
Drug: Medroxyprogesterone Acetate 500 MG — At a dosage of 500 mg/day
  Other Names: Medroxyprogesterone Acetate
  Arms: MA/MPA
Drug: Triprorelin Acetate — Intramuscular injection of 3.75mg was given 4 weeks apart and the maximum use are 6 courses
  Arms: GnRHa+letrozole
Drug: Letrozole 2.5mg — At a dosage of 2.5mg/day and no more than 24 weeks
  Other Names: Letrozole
  Arms: GnRHa+letrozole

SUMMARY:
To see if Gonadotropin-releasing hormone analogue (GnRHa) combined with aromatase inhibitors (AIs) will achieve better complete response rate than megestrol acetate or medroxyprogesterone acetate (MA/MPA) alone as fertility-sparing treatment for patients with early endometrial carcinoma.

DETAILED DESCRIPTION:
This will be a multicenter randomized controlled study to evaluate the treatment effects and adverse events of GnRHa plus AIs compared with MA/MPA in primary EEC patients.In this study, young patients (18-45 years) diagnosed as EEC for the first time seeking for fertility preserving treatment at the Obstetrics and Gynecology Hospital of Fudan University were screened. Patients were randomly assigned (1:1) to GnRHa+letrozole group (triprorelin acetate, intramuscular injection of 3.75mg was given 4 weeks apart and the maximum use are 6 courses. letrozole, 2.5mg oral daily and no more than 24 weeks) or MA/MPA group (160 mg oral MA daily or 500 mg oral MPA daily).

Hysteroscopy will be performed every 3 months during treatment to evaluate the treatment effects. For patients with EEC, complete response (CR) is defined as the reversion of endometrial carcinoma to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia with or without atypia; Stable disease (SD) is defined as the persistence of the disease; and progressive disease (PD) is defined as the progression of endometrial lesions. Continuous therapies will be needed in PR, SD or PD.The primary endpoint was cumulative complete response (CR) rate at 16 weeks of treatment. The secondary endpoints were cumulative CR rate at 28weeks of treatment, adverse events, recurrent rate, pregnancy rate, effects on ovarian function and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Consent informed and signed
* Primarily have a confirmed diagnosis of early-stage endometrial cancer (endometrioid, grade I, without myometrial inva- sion) ) based upon endometrial biopsy, diagnostic curettage or hysteroscopy
* No signs of suspicious myometrial invasion or extrauterine metastasis by enhanced magnetic resonance imaging (MRI), enhanced computed tomography (CT) or transvaginal ultrasonography (TVUS)
* Have a strong desire for remaining reproductive function or uterus
* Have good compliance and follow-up conditions, and patients are willing to follow up in Obstetrics and Gynecology Hospital of Fudan University in time

Exclusion Criteria:

* Pathologically confirmed as endometrial cancer with suspicious myometrial invasion or extrauterine metastasis
* Recurrent endometrial cancer
* Combined with severe medical disease or severely impaired liver and kidney function
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system; patients with breast cancer or other hormone- dependent tumors that cannot be used with progesterone
* Those who require hysterectomy or other methods other than conservative treatment with drugs
* Known or suspected pregnancy
* Contraindication for Medroxyprogesterone Acetate, Megestrol Acetate, Triprorelin Acetate, Letrozole or pregnancy
* Hormone treatment within 3 months before entering the trial;
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Complete response rates within 16 weeks of treatment | From date of treatment initiation until the date of CR, assessed up to 16 weeks.
  The cumulative 16-week CR rates will be calculated in two groups

SECONDARY OUTCOMES:
Complete response rates within 28 weeks of treatment | From date of treatment initiation until the date of CR, assessed up to 28 weeks.
  The cumulative 28-week CR rates will be calculated in two groups
Time to achieve complete response | From date of treatment initiation until the date of CR or date of hysterectomy,From date of randomization until the date of CR, assessed up to 2 years
  The median CR time will be calculated in two groups
Adverse events | From date of treatment initiation until the date of CR, assessed up to 2 years
  Adverse events related with Medroxyprogesterone Acetate, Megestrol Acetate, Triprorelin Acetate and Letrozole. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Quality of life during the treatment accessed by WHOQOL-BREF | From date of randomization until 12 weeks after treatment is over.
  Quality of life will be assessed at baseline, 4 weeks and every 12-16 weeks of treatment, using WHOQOL-BREF scale including assessment on pain, energy,sleep,mobil,activity,medication,work,positive feeling,think,esteem,body,negtivity,spirit,relationship,support,sex,safety,home,finance,service,information, environment,leisure,transport
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete response, they will be counted and the number of recurrence will be divided by number of patients followed up, then we can get the relapse rates. Comparison will be performed between two groups.
Change of AMH (anti-mullerian hormone ) serum level | From date of randomization until 24 weeks after treatment is over.
  AMH (anti-mullerian hormone ) will be assessed at baseline and every 12-16 weeks.
The rates of fertility outcomes | up to 2 years after the treatment for each patient
  The percentage of pregnancy and live-birth will be counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after this research being published,without patients personal information.
Supporting Information: Study Protocol
Time Frame: Data will be avaliable since this research being published
Access Criteria: Institutes or researchers who require the data should contact the principle investigator Prof.Xiaojun Chen via email that after this study being published.

REFERENCES:
- [Background] Zhou H, Cao D, Yang J, Shen K, Lang J. Gonadotropin-Releasing Hormone Agonist Combined With a Levonorgestrel-Releasing Intrauterine System or Letrozole for Fertility-Preserving Treatment of Endometrial Carcinoma and Complex Atypical Hyperplasia in Young Women. Int J Gynecol Cancer. 2017 Jul;27(6):1178-1182. doi: 10.1097/IGC.0000000000001008. PMID 28562472
- [Background] Rackow BW, Arici A. Endometrial cancer and fertility. Curr Opin Obstet Gynecol. 2006 Jun;18(3):245-52. doi: 10.1097/01.gco.0000193012.11523.c5. PMID 16735822
- [Background] Trimble CL, Kauderer J, Zaino R, Silverberg S, Lim PC, Burke JJ 2nd, Alberts D, Curtin J. Concurrent endometrial carcinoma in women with a biopsy diagnosis of atypical endometrial hyperplasia: a Gynecologic Oncology Group study. Cancer. 2006 Feb 15;106(4):812-9. doi: 10.1002/cncr.21650. PMID 16400639
- [Background] Corzo C, Barrientos Santillan N, Westin SN, Ramirez PT. Updates on Conservative Management of Endometrial Cancer. J Minim Invasive Gynecol. 2018 Feb;25(2):308-313. doi: 10.1016/j.jmig.2017.07.022. Epub 2017 Aug 3. PMID 28782618
- [Background] Gressel GM, Parkash V, Pal L. Management options and fertility-preserving therapy for premenopausal endometrial hyperplasia and early-stage endometrial cancer. Int J Gynaecol Obstet. 2015 Dec;131(3):234-9. doi: 10.1016/j.ijgo.2015.06.031. Epub 2015 Sep 8. PMID 26384790
- [Background] Baek JS, Lee WH, Kang WD, Kim SM. Fertility-preserving treatment in complex atypical hyperplasia and early endometrial cancer in young women with oral progestin: Is it effective? Obstet Gynecol Sci. 2016 Jan;59(1):24-31. doi: 10.5468/ogs.2016.59.1.24. Epub 2016 Jan 15. PMID 26866032
- [Background] Gunderson CC, Fader AN, Carson KA, Bristow RE. Oncologic and reproductive outcomes with progestin therapy in women with endometrial hyperplasia and grade 1 adenocarcinoma: a systematic review. Gynecol Oncol. 2012 May;125(2):477-82. doi: 10.1016/j.ygyno.2012.01.003. Epub 2012 Jan 11. PMID 22245711
- [Background] Chen M, Jin Y, Li Y, Bi Y, Shan Y, Pan L. Oncologic and reproductive outcomes after fertility-sparing management with oral progestin for women with complex endometrial hyperplasia and endometrial cancer. Int J Gynaecol Obstet. 2016 Jan;132(1):34-8. doi: 10.1016/j.ijgo.2015.06.046. Epub 2015 Oct 1. PMID 26493012
- [Background] Yang B, Xu Y, Zhu Q, Xie L, Shan W, Ning C, Xie B, Shi Y, Luo X, Zhang H, Chen X. Treatment efficiency of comprehensive hysteroscopic evaluation and lesion resection combined with progestin therapy in young women with endometrial atypical hyperplasia and endometrial cancer. Gynecol Oncol. 2019 Apr;153(1):55-62. doi: 10.1016/j.ygyno.2019.01.014. Epub 2019 Jan 21. PMID 30674421
- [Background] Mitsuhashi A, Habu Y, Kobayashi T, Kawarai Y, Ishikawa H, Usui H, Shozu M. Long-term outcomes of progestin plus metformin as a fertility-sparing treatment for atypical endometrial hyperplasia and endometrial cancer patients. J Gynecol Oncol. 2019 Nov;30(6):e90. doi: 10.3802/jgo.2019.30.e90. PMID 31576686
- [Background] Park JY, Kim DY, Kim JH, Kim YM, Kim KR, Kim YT, Seong SJ, Kim TJ, Kim JW, Kim SM, Bae DS, Nam JH. Long-term oncologic outcomes after fertility-sparing management using oral progestin for young women with endometrial cancer (KGOG 2002). Eur J Cancer. 2013 Mar;49(4):868-74. doi: 10.1016/j.ejca.2012.09.017. Epub 2012 Oct 13. PMID 23072814
- [Background] Ignatov A, Ortmann O. Endocrine Risk Factors of Endometrial Cancer: Polycystic Ovary Syndrome, Oral Contraceptives, Infertility, Tamoxifen. Cancers (Basel). 2020 Jul 2;12(7):1766. doi: 10.3390/cancers12071766. PMID 32630728
- [Background] Emons G, Schally AV. The use of luteinizing hormone releasing hormone agonists and antagonists in gynaecological cancers. Hum Reprod. 1994 Jul;9(7):1364-79. doi: 10.1093/oxfordjournals.humrep.a138714. PMID 7962452
- [Background] Grundker C, Volker P, Schulz KD, Emons G. Luteinizing hormone-releasing hormone agonist triptorelin and antagonist cetrorelix inhibit EGF-induced c-fos expression in human gynecological cancers. Gynecol Oncol. 2000 Aug;78(2):194-202. doi: 10.1006/gyno.2000.5863. PMID 10926802
- [Background] Grundker C, Emons G. The Role of Gonadotropin-Releasing Hormone in Cancer Cell Proliferation and Metastasis. Front Endocrinol (Lausanne). 2017 Aug 4;8:187. doi: 10.3389/fendo.2017.00187. eCollection 2017. PMID 28824547
- [Background] Azim A, Oktay K. Letrozole for ovulation induction and fertility preservation by embryo cryopreservation in young women with endometrial carcinoma. Fertil Steril. 2007 Sep;88(3):657-64. doi: 10.1016/j.fertnstert.2006.12.068. Epub 2007 Apr 10. PMID 17428480
- [Background] Barker LC, Brand IR, Crawford SM. Sustained effect of the aromatase inhibitors anastrozole and letrozole on endometrial thickness in patients with endometrial hyperplasia and endometrial carcinoma. Curr Med Res Opin. 2009 May;25(5):1105-9. doi: 10.1185/03007990902860549. PMID 19301987
- [Background] Minig L, Franchi D, Boveri S, Casadio C, Bocciolone L, Sideri M. Progestin intrauterine device and GnRH analogue for uterus-sparing treatment of endometrial precancers and well-differentiated early endometrial carcinoma in young women. Ann Oncol. 2011 Mar;22(3):643-649. doi: 10.1093/annonc/mdq463. Epub 2010 Sep 28. PMID 20876910
- [Background] Zhang Z, Huang H, Feng F, Wang J, Cheng N. A pilot study of gonadotropin-releasing hormone agonist combined with aromatase inhibitor as fertility-sparing treatment in obese patients with endometrial cancer. J Gynecol Oncol. 2019 Jul;30(4):e61. doi: 10.3802/jgo.2019.30.e61. Epub 2019 Feb 26. PMID 31074242
- [Background] Yin J, Ma S, Shan Y, Wang Y, Li Y, Jin Y, Pan L. Risk Factors for Recurrence in Patients with Atypical Endometrial Hyperplasia and Endometrioid Adenocarcinoma after Fertility-Sparing Treatments. Cancer Prev Res (Phila). 2020 Apr;13(4):403-410. doi: 10.1158/1940-6207.CAPR-19-0399. Epub 2020 Feb 3. PMID 32015095
- [Background] Tock S, Jadoul P, Squifflet JL, Marbaix E, Baurain JF, Luyckx M. Fertility Sparing Treatment in Patients With Early Stage Endometrial Cancer, Using a Combination of Surgery and GnRH Agonist: A Monocentric Retrospective Study and Review of the Literature. Front Med (Lausanne). 2018 Aug 27;5:240. doi: 10.3389/fmed.2018.00240. eCollection 2018. PMID 30211167
- [Background] McCaig FM, Renshaw L, Williams L, Young O, Murray J, Macaskill EJ, McHugh M, Hannon R, Dixon JM. A study of the effects of the aromatase inhibitors anastrozole and letrozole on bone metabolism in postmenopausal women with estrogen receptor-positive breast cancer. Breast Cancer Res Treat. 2010 Feb;119(3):643-51. doi: 10.1007/s10549-009-0646-0. PMID 19941160